CLINICAL TRIAL: NCT00004052
Title: Phase II, Multicenter Vaccination of Patients With Chronic Myelogenous Leukemia With a Multivalent Tumor Specific Breakpoint Peptide Vaccine
Brief Title: Vaccine Therapy in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-012; CDR0000067247 (Registry Identifier: PDQ (Physician Data Query)); NCI-H99-0036
Record Dates: First submitted 1999-12-10; First posted 2003-05-08 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — saponin QA-21V1

INTERVENTIONS:
Biological: QS21
Biological: bcr-abl peptide vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and immunogenicity of a multivalent tumor-specific breakpoint peptide vaccine in patients with chronic myelogenous leukemia.
* Determine the antileukemic effects of vaccination with these peptides in these patients.

OUTLINE: Patients receive bcr/abl breakpoint peptide vaccine in QS21 adjuvant subcutaneously at rotated sites every 1-3 weeks (on or about days 0, 7, 21, 35, and 56) over 8 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients demonstrating a response by week 10 may receive 3 additional monthly vaccinations initiated within 8 weeks of the fifth dose. Patients demonstrating a response by vaccination 8 may receive 3 additional vaccinations administered at two-month intervals.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven chronic myelogenous leukemia

  * Must have (9;22) translocation or bcr/abl transcript, and b3a2 breakpoint
  * No accelerated or blastic phase
* Must be in hematologic remission with peripheral WBC less than 20,000/mm^3

PATIENT CHARACTERISTICS:

Age:

* Over 16

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Absolute granulocyte count greater than 1,200/mm^3
* Platelet count greater than 70,000/mm^3
* Hemoglobin greater than 9.0 g/dL
* No active bleeding

Hepatic:

* Bilirubin less than 2.0 mg/dL
* Lactate dehydrogenase less than 2 times normal

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* No uncontrolled active infection requiring antibiotics
* No other serious illness
* No immunodeficiency other than from prior bone marrow transplantation
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 months since prior allogeneic or autologous bone marrow transplantation
* Prior vaccination with pentavalent peptide at less than study dose level allowed
* At least 4 weeks since prior immunotherapy other than interferon, donor lymphocyte infusion, or pentavalent vaccine
* Concurrent interferon allowed

Chemotherapy:

* At least 2 weeks since prior low-dose subcutaneous cytarabine
* At least 4 weeks since prior chemotherapy other than hydroxyurea
* No concurrent chemotherapy except hydroxyurea

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* No concurrent surgery

Other:

* Concurrent imatinib mesylate allowed
* No other concurrent systemic therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1999-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Cathcart, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas